CLINICAL TRIAL: NCT01234675
Title: The Effects of Milnacipran on Sleep Disturbance in Fibromyalgia
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Mansoor Ahmed M.D. (Other)
Collaborators: Forest Laboratories (Industry)
Responsible Party: Sponsor-Investigator, Mansoor Ahmed M.D., Medical Director, Cleveland Sleep Research Center
Organization: Cleveland Sleep Research Center (Other)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: SAV-MD-17
Record Dates: First submitted 2010-11-03; First posted 2010-11-04 (Estimated); Results first posted 2015-07-22 (Estimated); Last update posted 2019-08-21 (Actual); Status verified 2019-08

CONDITIONS: Sleep Disorders; Fibromyalgia; Sleep
Keywords: Fibromyalgia; Sleep disorders; Forest Laboratories; Milnacipran
MeSH Terms: conditions — Sleep Wake Disorders; Fibromyalgia | interventions — Milnacipran; Sugars

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- milnacipran (Experimental): Drug: milnacipran 7-day dose escalation, 28- day treatment with milnacipran 50 mg and 7-day taper period before or after crossover to placebo
  Interventions: Drug: Milnacipran
- placebo (Placebo Comparator): Drug: placebo 45-day placebo treatment before or after crossover to milnacipran
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Milnacipran — 50 mg twice daily
  Other Names: Savella
  Arms: milnacipran
Drug: Placebo — 50 mg twice daily
  Other Names: Sugar pill
  Arms: placebo

SUMMARY:
Fibromyalgia is a condition of chronic widespread pain, sleep disturbance and fatigue. Most of the patients with fibromyalgia complain of either non-restorative sleep or complaints of disturbed sleep due to pain. The study aimed at examining the effects of milnacipran on sleep disturbance in patients with fibromyalgia. The study is a randomized, double-blind, placebo controlled, two way crossover polysomnography (PSG) study to explore the effects of milnacipran on sleep disturbance. Patients received either milnacipran 50 mg twice a day (BID) or matching placebo.

DETAILED DESCRIPTION:
The sleep disturbance in fibromyalgia is characterized as non-restorative in nature, and is defined as a feeling of light sleep, independent of duration, and as non-refreshing. As such, these patients wake up in the morning and complain of stiffness and overall aching of the body.

It is well known that reciprocal relationship exists between sleep and pain, with sleep disturbances being an important contributor to morbidity in fibromyalgia. Milnacipran, a selective serotonin norepinephrine receptor inhibitor (SNRI), was approved by the Food and Drug Administration (FDA) for the management of fibromyalgia. Although milnacipran has extensively been studied in fibromyalgia patients, but there is no objective measure, i.e., the use of overnight polysomnography, to determine its effects on sleep.

The study was undertaken to evaluate the effects of milnacipran on PSG determined measures of sleep in patients with fibromyalgia. The study also evaluated the impact of milnacipran on subjective measures of sleep and fibromyalgia symptoms.

ELIGIBILITY:
Inclusion Criteria:

1. Men or women at least 18 years or older
2. Diagnosis of fibromyalgia
3. Clinically significant sleep disturbance, defined as difficulty in maintaining sleep (wake after sleep onset and arousal index) at least three times per week for at least one month
4. Understand and willing to cooperate with the study procedures
5. Maintain a normal sleep schedule, with daytime-awake and nighttime-sleep schedule, with customary bedtime between 9 PM and midnight, and rise time 5 AM and 9 AM
6. Patients who are able to speak, read, and understand English language and able to follow the study protocol, and are able to sign the informed consent

Exclusion Criteria:

1. Subject has any of the following medical conditions:

   Liver disease, blood disorder, autoimmune disease, endocrine, cardiovascular, hypertension, renal, hepatic, gastrointestinal, or neurological disorder, active peptic ulcer or inflammatory bowel disease
2. Significant sleep apnea
3. Periodic leg movement disorder (PLMD) or restless legs syndrome (RLS)
4. Any form of severe psychiatric illness, moderate to severe depression, including significant risk of suicide
5. Patients with uncontrolled glaucoma
6. Inability to discontinue the prohibited medications
7. Female of childbearing potential not using birth control measures; or lactating.
8. History of alcohol, narcotic, benzodiazepines or other substance abuse within the past one year.
9. Patient on prohibited medication will include but not limited to:

   * Anxiolytics, anti-convulsants, antipsychotics, lithium, barbiturates, anti-histamines, monoamine oxidase inhibitors, or medications that affect sleep
   * Any prescription or over the counter stimulants
   * Medications that are contraindicated with the use of milnacipran
10. Excessive caffeine use, defined as a consumption of more than 500 mg of caffeine or other xanthines, smoking >1/2 a pack/day or alcohol use >14 units/week
11. History of allergy to milnacipran.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2010-11; Primary Completion 2014-02 (Actual); Study Completion 2014-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mansoor Ahmed, MD, Principal Investigator — Cleveland Sleep Research Cneter; Rozina Aamir, MS, MBA, Study Director — Cleveland Sleep Research Center; Noel Cyrill, MD, Study Director — SouthWest Cleveland Sleep Center; Nosson S Goldfarb, M.D., Study Director — Cleveland Sleep Research Center
Locations (1):
- Cleveland Sleep Research Center, Middleburg Heights, Ohio, United States

REFERENCES:
- [Derived] Ahmed M, Aamir R, Jishi Z, Scharf MB. The Effects of Milnacipran on Sleep Disturbance in Fibromyalgia: A Randomized, Double-Blind, Placebo-Controlled, Two-Way Crossover Study. J Clin Sleep Med. 2016 Jan;12(1):79-86. doi: 10.5664/jcsm.5400. PMID 26414990

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo Then Milnacipran; Milnacipran Then Placebo: 50 mg twice daily (BID) maintenance dose
Period: First Intervention (6 Weeks)
Arm/Group | Placebo Then Milnacipran | Milnacipran Then Placebo
Started | 10 | 9
Completed | 9 | 8
Not Completed | 1 | 1
Not completed — Adverse Event | 0 | 1
Not completed — Withdrawal by Subject | 1 | 0
Period: Second Intervention (6 Weeks)
Arm/Group | Placebo Then Milnacipran | Milnacipran Then Placebo
Started | 9 | 8
Completed | 7 | 8
Not Completed | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- All Study Participants: 2 treatment period, with each period 6 weeks and 7 day washout period Milnacipran in treatment period 1, Placebo in treatment period 2 Placebo treatment in Period 1, and Milnacipran in Period 2
Arm/Group | All Study Participants
Number analyzed (Participants) | 19
Age, Continuous [Mean (Full Range); unit: years] | 49.2 [28 to 72]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17
  Male | 2
Baseline polysomnographic sleep parameters [Mean (Standard Deviation); unit: minutes]
  Latency to persistent sleep (LPS) | 49.4 (43.4)
  Total sleep time (TST) | 340.7 (78.9)
  Wake after sleep onset (WASO) | 97.2 (70.6)
Number of awakenings after sleep onset (NAASO) [Mean (Standard Deviation); unit: awakenings] | 31.9 (12.9)
Sleep efficiency (SE) [Mean (Standard Deviation); unit: percentage of total sleep time] | 72.3 (15.8)
Arousal index (AI) [Mean (Standard Deviation); unit: arousals per hour] | 24.8 (9.8)
Total stage shifts [Mean (Standard Deviation); unit: Stage shifts] — Sleep stage shifts: stage 1, stage 2, stage 3, REM sleep
  Stage shifts | 147.4 (42.2)
Rapid Eye Movement (REM) latency [Mean (Standard Deviation); unit: minutes] — Time from sleep onset to the first epoch of rapid eye movement (REM) sleep
  minutes | 126.5 (91.3)
Sleep architecture [Mean (Standard Deviation); unit: percentage of total sleep time] — Pattern of sleep as it shifts between the different sleep stages. Sleep stages 1-3 are collectively referred to as non--rapid eye movement sleep (NREM)
  percentage of total sleep time
    Stage N1 | 18.9 (6.6)
    Stage N2 | 59.0 (13)
    Stage N3 | 4.2 (8.4)
    REM Sleep | 18.0 (7.3)

OUTCOME MEASURES:

1. Primary Outcome: Number of Awakenings After Sleep Onset (NAASO)
Description: Number of awakenings after defined sleep onset until lights on.
Time Frame: 4-Week maintenance treatment with milnacipran and placebo
Population: 15 subjects completed the study
Measure: Mean (Standard Error); unit: Awakenings
Groups:
- Milnacipran: Treatment with 50 mg BiD
- Placebo: 50 mg placebo BiD
Arm/Group | Milnacipran | Placebo
Number analyzed (Participants) | 15 | 15
Awakenings | 39.5 (4.5) | 34.9 (4.2)
Statistical Analysis 1: Comparison: Milnacipran vs Placebo; Test type: Superiority; p = 0.424, Paired T test; Paired difference = 4.6, 95% CI 2-sided [-7.3 to 16.6]

2. Primary Outcome: Sleep Efficiency (SE)
Description: Percentage of time spent asleep while in bed
Time Frame: 4-Week maintenance treatment with milnacipran and placebo
Measure: Mean (Standard Error); unit: percentage of total sleep time
Arm/Group | Milnacipran | Placebo
Number analyzed (Participants) | 15 | 15
percentage of total sleep time | 77.1 (3.8) | 83.3 (2.3)
Statistical Analysis 1: Comparison: Milnacipran; Test type: Superiority; p = 0.049, Paired T test; Paired difference = -6.1, 95% CI 2-sided [-12.2 to -0.04]

3. Primary Outcome: Wake After Sleep Onset (WASO)
Description: Wake time after defined sleep onset until lights on.
Time Frame: 4-Week maintenance treatment with milnacipran and placebo
Measure: Mean (Standard Error); unit: minutes
Arm/Group | Milnacipran | Placebo
Number analyzed (Participants) | 15 | 15
minutes | 76.2 (10.8) | 53.6 (8.1)
Statistical Analysis 1: Comparison: Milnacipran vs Placebo; Test type: Superiority; p = 0.056, Paired T test; Paired difference = 22.6, 95% CI 2-sided [-0.6 to 45.8]

4. Secondary Outcome: Latency to Persistent Sleep Onset (LPS)
Description: It is defined as time from lights out to the first consecutive 2 minutes of uninterrupted sleep.
Time Frame: 4-Week treatment with milnacipran and placebo
Measure: Mean (Standard Error); unit: minutes
Arm/Group | Milnacipran | Placebo
Number analyzed (Participants) | 15 | 15
minutes | 41.6 (6.2) | 38.6 (5.8)
Statistical Analysis 1: Comparison: Milnacipran vs Placebo; Test type: Superiority; p = 0.683, Paired T test; Paired difference = -6.1, 95% CI 2-sided [-12.5 to 18.5]

5. Secondary Outcome: Total Sleep Time (TST)
Description: Total sleep of all Rapid Eye Movement (REM) and Non- Rapid Eye Movement Sleep (NTREM) from lights out to lights on.
Time Frame: 4-Week treatment with milnacipran and placebo
Measure: Mean (Standard Error); unit: minutes
Arm/Group | Milnacipran | Placebo
Number analyzed (Participants) | 15 | 15
minutes | 361.7 (19.6) | 386.1 (12.5)
Statistical Analysis 1: Comparison: Milnacipran vs Placebo; Test type: Superiority; p = 0.155, Paired T test; Paired difference = -1.502, 95% CI 2-sided [-59.1 to 10.4]

6. Secondary Outcome: Arousal Index (AI)
Description: Number of arousals per hour of sleep
Time Frame: 4-Week treatment with milnacipran and placebo
Measure: Mean (Standard Error); unit: arousals per hour
Arm/Group | Milnacipran | Placebo
Number analyzed (Participants) | 15 | 15
arousals per hour | 30.2 (2.2) | 31.2 (4.0)
Statistical Analysis 1: Comparison: Milnacipran vs Placebo; Test type: Superiority; p = 0.805, Paired T test; Paired difference = -1.0, 95% CI 2-sided [-9.8 to 7.8]

7. Secondary Outcome: Slow Wave Sleep (SWS)
Description: Time spent in stage 3 of non-rapid eye movement sleep and often referred to as deep sleep.
Time Frame: 4-Week treatment with milnacipran and placebo
Measure: Mean (Standard Error); unit: percentage of total sleep time
Arm/Group | Milnacipran | Placebo
Number analyzed (Participants) | 15 | 15
percentage of total sleep time | 8.4 (2.7) | 9.4 (2.6)
Statistical Analysis 1: Comparison: Milnacipran vs Placebo; Test type: Superiority; p = 0.844, Paired T test; Paired difference = -1.0, 95% CI 2-sided [-11.6 to 9.6]

8. Secondary Outcome: Sleep Problem Index 2, Medical Outcomes Study Sleep Scale (MOS-SS)
Description: This is a subjective index derived from the medical outcomes study sleep scale (MOS-SS) scored on a 0-100 possible range with higher scores indicating more severe sleep disruption. The scale is a self-report instrument consisting of 12 items that assess perceived initiation and maintenance of sleep, respiratory problems during sleep, sleep duration, perceived adequacy of sleep and daytime somnolence.
Time Frame: 4-Week treatment with milnacipran and placebo
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Milnacipran | Placebo
Number analyzed (Participants) | 15 | 15
score on a scale | 37.8 (4.4) | 34.9 (3.8)
Statistical Analysis 1: Comparison: Milnacipran vs Placebo; Test type: Superiority; p = 0.509, Paired T test; Paired difference = 2.9, 95% CI 2-sided [-6.4 to 12.2]

9. Secondary Outcome: Sleep Quality Scale
Description: Sleep quality measure derived from daily sleep diary rating ranging from 0 ("very poor") to 10 ("excellent")
Time Frame: 4-Week treatment with milnacipran and placebo
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Milnacipran | Placebo
Number analyzed (Participants) | 15 | 15
score on a scale | 5.2 (0.52) | 4.9 (0.4)
Statistical Analysis 1: Comparison: Milnacipran vs Placebo; Test type: Superiority; p = 0.3, Paired T test; Paired difference = 0.32, 95% CI 2-sided [-0.3 to 0.6]

10. Secondary Outcome: Fatigue Severity Scale (FSS) Total Score
Description: The scale is a 9-item self-report of fatigue in the past week and scored on a 7-point scale with 1 = strongly disagree and 7 = strongly agree. Scores range from 9 to 63 with higher scores indicating higher fatigue severity. A total score greater or equal to 36 suggests fatigue.
Time Frame: 4-Week treatment with milnacipran and placebo
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Milnacipran | Placebo
Number analyzed (Participants) | 15 | 15
score on a scale | 41.0 (3.4) | 42.3 (3.1)
Statistical Analysis 1: Comparison: Milnacipran vs Placebo; Test type: Superiority; p = 0.685, Paired T test; Paired difference = -1.03, 95% CI 2-sided [-8.2 to 5.6]

11. Secondary Outcome: Fibromyalgia Impact Questionnaire (FIQ) Total Score
Description: The scale is composed of 10 items relating to fibromyalgia symptoms experienced in the past week. Score ranges from 0 to 100 with higher scores indicating a greater effect of fibromyalgia on a person's life.
Time Frame: 4-Week treatment with milnacipran and placebo
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Milnacipran | Placebo
Number analyzed (Participants) | 15 | 15
score on a scale | 40.0 (6.8) | 45.3 (4.0)
Statistical Analysis 1: Comparison: Milnacipran vs Placebo; Test type: Superiority; p = 0.349, Paired T test; Paired difference = -5.3, 95% CI 2-sided [-17.0 to 6.4]

12. Secondary Outcome: Brief Pain Inventory (BPI) Mean Severity Score
Description: The score is derived from the BPI scale and measures pain intensity in the past 24 hour. The pain severity score is derived as the average score of 4 pain items assessing pain at its "worst", "least", "average" and "now" and ranges from 0-10 with higher scores reflecting greater pain
Time Frame: 4-Week treatment with milnacipran and placebo
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Milnacipran | Placebo
Number analyzed (Participants) | 15 | 15
score on a scale | 4.1 (0.6) | 4.7 (0.4)
Statistical Analysis 1: Comparison: Milnacipran vs Placebo; Test type: Superiority; p = 0.305, Paired T test; Paired difference = -0.6, 95% CI 2-sided [-1.8 to 5.6]

13. Secondary Outcome: Brief Pain Inventory (BPI) Mean Interference Score
Description: The score is derived from the BPI scale and measures the effect of pain on functioning in the past 24 hour. It is the average score of 7 items interfering with general activity, mood, walking ability, normal work, relations with other people, sleep and enjoyment of life. Score ranges from 0-10 with higher scores reflecting greater interference.
Time Frame: 4-Week treatment with milnacipran and placebo
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Milnacipran | Placebo
Number analyzed (Participants) | 15 | 15
score on a scale | 3.8 (0.6) | 4.3 (0.5)
Statistical Analysis 1: Comparison: Milnacipran vs Placebo; Test type: Superiority; p = 0.425, Paired T test; Paired difference = -0.5, 95% CI 2-sided [-1.8 to 0.8]

ADVERSE EVENTS:
Time Frame: Adverse event data was collected on and after Day 1 of the first treatment period. The data collection continued till the two weeks after the second treatment period.
Description: Additional data was collected after the end of study visit if the patient reported an adverse event.
Groups:
- Milnacipran: Drug: milnacipran, 50 mg twice daily for 4 weeks.
- Placebo: Drug: Placebo 50 mg, twice daily for 4 weeks.
Arm/Group | Milnacipran | Placebo
Serious Adverse Events (participants affected / at risk) | 0/19 | 1/19
Other Adverse Events (participants affected / at risk) | 12/19 | 10/19
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Milnacipran (N=19) | Placebo (N=19)
Gall Stones (Gastrointestinal disorders) | 0 (0) | 1 (1) — During the study the subject was diagnosed with having gall stones. After the blind was broken, the site found out that she was on placebo, and was never treated with the study drug.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Milnacipran (N=19) | Placebo (N=19)
nausea (Gastrointestinal disorders) | 4 (4) | 0 (0) — nausea and vomiting
Headache (Nervous system disorders) | 3 (3) | 0
Dry Mouth (General disorders) | 1 (1) | 1 (1)
Flushing (Nervous system disorders) | 2 (2) | 0 (0)
Constipation (Gastrointestinal disorders) | 2 (2) | 2 (2)
Abdominal pain (Gastrointestinal disorders) | 2 (2) | 3 (3)
Sinusitis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Worsening of pain (Nervous system disorders) | 0 (0) | 2 (2)
Increased Perspirations (General disorders) | 1 (1) | 0 (0)
cold/flu (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Increased Heartrate (Cardiac disorders) | 1 (1) | 0 (0)
diarrhea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Excessive menstrual bleeding (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Streptococcal infection (throat) (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Excessive urination (Renal and urinary disorders) | 1 (1) | 0 (0)
Periodontal disease (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Elevated Blood Pressure (Cardiac disorders) | 0 (0) | 1 (1)
Cold sweats (General disorders) | 1 (1) | 0 (0)
Abnormal ejaculation (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Foot sprain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Pruritis (Immune system disorders) | 1 (1) | 0 (0)
Petechial rash (Immune system disorders) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
A well-established adaptation and re-adaptation to laboratory effects may have compromised our results. Other study biases include biases inherent in the crossover design, and a small sample size.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No